CLINICAL TRIAL: NCT04672616
Title: Inklusiv Plus: Mental Health Of Unemployed Adolescents And Young Adults
Acronym: Ip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zurich University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Filomena Sabatella, Prinicipal Investigator, Zurich University of Applied Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020-02184
Record Dates: First submitted 2020-11-17; First posted 2020-12-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Mental Disorder
Keywords: emerging adulthood; unemployment; transition
MeSH Terms: conditions — Mental Disorders | interventions — Psychotherapy, Group

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group psychotherapy (Experimental): Weekly group meeting w/psychotherapist: All the participants fulfilling the eligibility criteria are asked to take part in an additional Intervention. The Intervention is a weekly group Meeting with a psychotherapist to discuss issues or problems the group members have
  Interventions: Behavioral: Group psychotherapy

INTERVENTIONS:
Behavioral: Group psychotherapy — The intervention is a group psychotherapeutic offer for mentally burdened adolescents and young adults to support their professional integration.

SUMMARY:
The expansion project "Inclusive Plus", which is financed by Innosuisse, is based on a pilot project. The psychotherapeutic offer developed in the previous project for psychologically burdened adolescents and young adults to support them in their professional integration was revised and supplemented and is being reviewed in this project. In addition to the group psychotherapeutic intervention, 5 one-on-one interviews are offered as needed. In addition, regular further training courses on mental health and illness in adolescence are implemented. And finally, a conference is to promote cooperation between referring physicians and bridge offers. The intervention will be implemented in 5 cantons (Zurich, Berne, Lucerne, St. Gallen, Appenzell Ausserrhoden) and in 7 different bridge services. The program is aimed at adolescents and young adults between 16 and 29 years of age who have sufficient knowledge of German. Participation is voluntary and the group size for the psychotherapy group is limited to 8 participants. The main question is whether the integration of young people with mental stress into the labor market is more successful. At three points in time (entry, exit, six months after exit) changes in selected indicators (including work ability, mental health, functional status, behaviour in seeking help) are measured. In addition, changes in the groups of participants will be surveyed. The implementation of the psychotherapy groups in the respective bridge offers will take place in autumn 2020, and the study will be completed with the last follow-up by the end of 2022.

DETAILED DESCRIPTION:
In Switzerland, almost one in six young people has no further professional solution after the compulsory school years. So-called bridge offers have been created for these young people. Despite these offers, adolescents and young adults with multiple burdens often do not find a training place or job. Young people who have not found a follow-up solution are significantly more likely to suffer from mental impairments and disorders than those who begin an apprenticeship or attend secondary school. According to Sabatella and von Wyl, this may be due on the one hand to the fact that a lack of an apprenticeship places a psychological burden on them. On the other hand, it can be assumed that many young people do not find an apprenticeship or job precisely because of a mental illness. Furthermore, the psychological impairments and illnesses are often not recognized or treated. This is probably due to the fact that young people often fail to make use of appropriate psychotherapeutic services, on the one hand because of the fear of being stigmatized, and on the other hand because they often seem to lack the insight to need and make use of help. The problem of mental stress and illness in adolescence is also reflected in IV consultations. The rate of new pensioners is significantly higher among 18 to 19-year-olds. Early treatment without delay can positively influence the course of an illness. In contrast, it has been shown that the longer people wait to treat a mental illness, the greater the risk of chronification. Therefore, treatment of mental illness is especially important for young people. The further development of these young people is not - as often feared - impaired. On the contrary, their professional and personal future prospects become more positive. As a result, cases of full retirement can be reduced, which has a positive effect on health costs.

Against this background, the pilot project "inclusive", which preceded this project and was financed by the Gebert Rüf Foundation, was carried out. In cooperation with the bridge offer lifetime health, an innovative approach for a better integration of work was developed, applied and tested for two years: The existing care team of lifetime health was supplemented by a psychotherapist who conducted a 90-minute weekly group psychotherapy session with the young clients of lifetime health. He was also in contact with the team and the clients as needed.

This (group) psychotherapeutic offer developed in the previous project for mentally burdened adolescents and young adults to support them in their professional integration was revised and supplemented. In the current project phase it is being implemented in 7 further bridge offers in five cantons. For an initial assessment of whether such an offer is also suitable for adults, a group is also offered for adults at one of the locations. The project is financed by Innosuisse.

ELIGIBILITY:
Inclusion Criteria:

* Participation in work integration programme

Exclusion Criteria:

* Insufficient knowledge of German
* Participant is under guardianship which doesn't allow legal capacity to act

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Social functioning status | Up to 2 years
  The social functioning status is assessed using the Mini-ICF-APP (Linden et al., 2009), based on the International Classification of Functioning, Disability and Health (ICF) published by the WHO. The ICF is a complex document and the Mini-ICFAPP (Mini-ICF-Rating for limitations of Activities and Participation in Psychological disorders) was developed to allow the reliable and rapid measurement and recording of impairments of capacity. It is used in this study as a self-assessment tool to describe and quantify activity and participation impairments in the context of mental illness. 13 areas are rated on a five-point Likert-scale (0 =no impairment, 1 =mild impairment, 2 =moderate disability, 3 = severe disability, 4 =total disability). The self-rating scores will then be averaged in order to have one overall score and then this overall score will be compared on three different time points (pre-treatment, post treatment and 6 months follow up). High scores here mean high impairment.

SECONDARY OUTCOMES:
Change in Work Ability | Up to 2 years
  The Work Ability Index (WAI) is an instrument used in occupational health care and research to assess work ability of workers. The purpose of WAI is to help define necessary actions to maintain and promote work ability. The scoring system of the questionnaire categorises work ability, with recommendations for action provided for each category. Appropriate action can then be taken to prevent declining work ability. Each answer has a different score, with users calculating their total points to determine their final score. The minimum is 7, the maximum is 49. The four categories of scores and the objectives of the measures to be taken are as follows: 7-27 points (bad) - restore work ability; 28-36 points (moderate) - improve work ability; 37-43 points (good) - support work ability; 44-49 points (very good) - support work ability. This overall score will be compared on three different time points (pre-treatment, post treatment and 6 month follow up).

OTHER OUTCOMES:
Psychopathological symptoms | Up to 2 years
  Psychopathological symptoms are measured using the Brief Symptom Checklist (BSCL; Franke, 2000). The BSCL records any subjective impairment caused by physical and especially psychological symptoms The BSCL consists of 53 items, i.e. statements to which the patient is to say whether they apply not at all, a little, moderately, strongly or very strongly (not at all = 0, very strongly = 4). Higher values indicate greater stress. The psychological stress is recorded on nine scales (aggressiveness/ hostility, anxiety, depression, paranoid thinking, phobic anxiety, psychoticism, somatization, insecurity in social contact, compulsiveness) and three global parameters.
Structural impairments | Up to 2 years
  With the Operationalized Psychodynamic Diagnostics Structural Questionnaire (OPD-SFK; Ehrenthal et al., 2015) structural limitations of personality can be quickly mapped in the self-assessment with 12 items. The questions are answered according on a Likert scale: 0=not at all true, 1=rather not true, 2=partly true, 3=rather true, 4=totally true. The Self-perception subscale links aspects of the self with structural skills of emotion regulation, the Contact Shaping subscale links interactional skills with aspects of self-uncertainty. The Relationship Model subscale maps the representation of relationship experiences, associated with corresponding expectations for new relationships. The value range of the sum score is from 0 (="highest structural level") to 48 (="lowest structural level").
Interpersonal problems | Up to 2 years
  Interpersonal difficulties are recorded with the Inventory of Interpersonal Problems (IIP-D; Horowitz et al., 2016). The scale comprises 32 items. The IIP identifies respondents as "hard to do" (i.e., behavioral inhibitions) or "does too much" (i.e., behavioral excesses) on a 0 (not at all) to 4 (extremely) Likert-type scale. It provides an overall score and 8 subscale scores: domineering, vindictive, cold, socially avoidant, non-assertive, exploitable, overly nurturant, and intrusive. The overall score shows the extent of interpersonal problems.

CONTACTS AND LOCATIONS:
Overall Officials: Agnes von Wyl, Prof, Principal Investigator — University of applied sciences
Locations (1):
- ZHAW, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No